CLINICAL TRIAL: NCT03848611
Title: Combination of CM082 With JS001 in Patients With Advanced Non-Small Cell Lung Cancer (SCLC) Who Progressed on First-line Treatment: a Phase II Study
Brief Title: CM082 and JS001 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AnewPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM082-CA-IV-401
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vorolanib; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM082 plus JS001 (Experimental): Patients who meet the enrollment criteria will receive CM082 tablets 150mg once daily (qd) orally (taken within half an hour after daily breakfast) in combination with JS001 (3mg/kg, once every 2 weeks, q2w), every 28 days A treatment cycle until the disease progresses, the toxicity is intolerable, the investigator or subject decides to withdraw, loses to follow up, starts using other anti-tumor treatments or dies.
  Interventions: Drug: CM082 plus JS001

INTERVENTIONS:
Drug: CM082 plus JS001 — CM082：150mg once a day (qd) orally (taken within half an hour after breakfast). JS001 :An intravenous infusion of a solution having a concentration of 1-10 mg/ml was prepared with 0.9% physiological saline, and administered once every two weeks. Using an inline filter (0.2 or 0.22 μm), the drug was diluted with physiological saline and intravenously administered within 60 minutes.
  Other Names: Vorolanib plus Toripalimab Injection

SUMMARY:
This study was a one-arm, single-center, phase II clinical study. Patients who meet the enrollment criteria will receive CM082 tablets 150mg once daily (qd) orally (taken within half an hour after daily breakfast) in combination with JS001 (3mg/kg, once every 2 weeks, q2w), every 28 days a treatment cycle until the disease progresses, the toxicity is intolerable, the investigator or subject decides to withdraw, loses to follow up, starts using other anti-tumor treatments or dies.

DETAILED DESCRIPTION:
The study is divided into the following five stages--screening period, treatment period, end of treatment / withdrawal treatment, follow-up after treatment, survival follow-up.

Screening period Subjects should be informed and signed an informed consent form prior to screening assessment. Screening should be performed within 28 days prior to dosing. After the investigator confirms compliance with the inclusion criteria and does not meet the exclusion criteria, the subject may be enrolled in the study drug.

Treatment period At this stage the subject will be treated with CM082 and JS001 until disease progression, intolerable toxicity, the investigator or subject decides to quit, is lost to follow-up, begins using other anti-tumor treatments or dies.

During the trial, subjects received a safety assessment every 4 weeks; tumor assessments were performed 6 weeks after the first visit and every 8 weeks after the first tumor assessment. Tumor progression will be evaluated simultaneously according to RECIST criteria and iRECIST criteria. Subjects identified as confirmed progressive disease(iCPD) according to iRECIST criteria should discontinue treatment.

End of treatment / withdrawal treatment End of treatment(EOT)visit evaluation should be performed as soon as possible after the subject has discontinued the test drug. Anyone who discontinues treatment or withdraws from treatment for reasons other than progression of the disease should perform a safety assessment as soon as possible, while continuing to perform a tumor assessment at the same frequency as the treatment period until disease progression or initiation of other anti-tumor treatments. However, subjects who have terminated treatment due to disease progression need only undergo a safety assessment and no longer have a tumor assessment. If the subject terminates treatment due to toxicity or other reasons at the last visit and does not continue taking the test drug afterwards, the visit is considered to be the end of treatment/exit treatment visit.

Follow-up after treatment For subjects who completed the trial or withdrew their informed consent, all adverse events (AEs) and concomitant medications must be recorded up to 30 days after the last dose of the trial, and all new AEs were issued within 30 days of the last trial dose. For subjects who started using other anti-tumor therapies, AEs that were not severe and that the investigator considered unrelated to the test drug were no longer recorded.

Survival follow-up Subjects with disease progression or other anti-tumor treatments will no longer undergo safety and tumor assessment, but continue to collect data on overall survival and follow-up treatment at telephone follow-up every 12 weeks until the patient dies or loses visit.

Note: Patients who discontinue treatment due to disease progression (except for patients withdrawing informed consent, loss of follow-up, death) should continue to follow the tumor assessments according to the original frequency (no safety assessment). Once disease progression has occurred or other anti-tumor drugs have been used, a telephone survival follow-up is performed every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of recurrence after surgery, inoperable resection or metastasis advanced NSCLC (III/IV period), with no specific driver gene mutations (EGFR or ALK).
* Has not received any systemic anti-tumor medication or adjust the chemotherapy regimen because of intolerance( but the treatment should be completed for at least 4 weeks prior to the first dose of study drug, and all related toxicity events have returned to normal or no more than Grade I of CTCAE 4.03, except for hair loss).
* Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1.
* Life expectancy of at least 12 weeks.
* All patients are suggested tumor tissue specimens (preferably fresh tissue specimens) for PD-L1 expression analysis prior to enrollment. If the subject did not undergo a pathological examination before participating in the trial, the collected tumor tissue specimens will also be used for pathological examination to confirm the diagnosis of NSCLC.
* There is at least one measurable lesion according to the RECIST 1.1 standard and the lesion has not received radiotherapy.
* Patients may have a history of brain/meningeal metastases, but must undergo topical treatment (surgery/radiotherapy) and be clinically stable for at least 3 months prior to the start of the study .If corticosteroids have been used before, they should be discontinued for at least 2 weeks before the first dose of study drug.
* The level of organ function must meet the following requirements (7 days before the first dose of study drug):

  * Bone marrow: Absolute neutrophil count (ANC) ≥ 1.5 × 109 / L, platelet (PLT) ≥ 100 × 109 / L, hemoglobin (HB) ≥ 9g / dL (no blood transfusion or receiving blood components within 14 days before detection);
  * Liver: serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal（ULN）, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5*ULN (if liver metastasis, AST, ALT allowed) ≤ 5 *ULN);
  * Serum creatinine ≤ 1.5*ULN and endogenous creatinine clearance ≥ 50milliliter(ml) / min (Cockcroft-Gault formula);
  * Well-controlled hypertensive patients can be enrolled;
  * International normalized ratio (INR), activated partial thromboplastin time (aPTT) ≤ 1.5 *ULN for patients who have not received anticoagulant therapy; patients who receive anticoagulant therapy should be treated within the requirements of label
  * Urine protein ≤ 1+, if urine protein > 1+, 24 hours urine protein measurement is required, the total amount of which needs ≤ 1 gram;
  * Free Triiodothyronine(FT3), Free Thyroxine(FT4), Thyroid-Stimulating Hormone(TSH) normal or abnormal has no clinical significance;
  * The heart function is normal, that is, the electrocardiogram is normal or abnormal has no clinical significance. The echocardiography shows that the left ventricular ejection fraction (LVEF) is greater than 50%.
* Serum pregnancy test results must be negative within 7 days prior to the first dose of the test drug for women of childbearing age; males with fertility or women who are at risk of pregnancy must use highly effective methods of contraception throughout the trial (eg oral contraceptives, intrauterine contraceptive device, controlled libido or barrier contraceptive method combined with spermicide), and continued contraception for 12 months after the end of treatment.
* Ability to understand the nature of this trial and give written informed consent. Willingness and ability to comply with trial and follow-up procedures.

Exclusion Criteria:

* Patients who have previously received anti-PD-1, anti-PD-L1, anti-PD-L2 therapy, or VEGFR Tyrosine Kinase Inhibitors(TKI) therapy.
* Patients currently receiving anti-tumor treatment.
* Patients who received large surgery within 4 weeks before the first dose of the test drug or has not recovered from the side effects of this operation, received live vaccination or immunotherapy within 4 weeks before the first dose of the test drug, and radiotherapy was performed within 2 weeks.
* Subjects with a history of malignancy (unless NSCLC) were excluded unless complete remission was achieved at least 2 years prior to enrollment and no further treatment was required during the study period (the following conditions are not limited: non-melanoma skin cancer) , bladder carcinoma in situ, gastric carcinoma in situ, colonic carcinoma in situ, endometrial carcinoma in situ, cervical carcinoma in situ/dysplasia, melanoma carcinoma in situ or breast carcinoma in situ)
* Hematopoietic stimulating factors were received within 1 week prior to the first dose of the study drug, such as granulocyte colony-stimulating factor (G-CSF) and erythropoietin.
* HIV antibody or Treponema pallidum antibody test results are positive.
* If HBsAg or HBcAb is positive, hepatitis B virus(HBV) DNA should be tested. Patients should be excluded if the measurement is above the upper limit of the normal range. If HCV antibody is positive, hepatitis C virus(HCV) DNA should be tested. Patients should be excluded if the measurement is above the upper limit of the normal range.
* Those known to be allergic to recombinant humanized PD-1 monoclonal antibody drugs and their components; those known to be allergic to CM082 and any of its excipients.
* A large amount of pleural or ascites with clinical symptoms and requiring symptomatic treatment.
* Active lung disease (eg, interstitial pneumonia, pneumonia, obstructive pulmonary disease, asthma) or a history of active tuberculosis.
* Have any clinical problems out of control, including but not limited to:

  * Persistent or active (severe) infection;
  * Hypertension that is not effectively controlled (blood pressure lasts greater than 150/90mmHg);
  * Diabetes that is not effectively controlled;
  * Heart disease, defined as grade III/IV congestive heart failure or heart block defined by the New York Heart Association
  * Having a history of or suspected of having an autoimmune disease;Having a history of any kind of disease requiring treatment with a steroid or immunosuppressive, such as: pituitary inflammation, colitis, hepatitis, nephritis, hyperthyroidism, Hypothyroidism, etc.;
  * The following situation occurred within 6 months before the first dose:

    * Deep vein thrombosis or pulmonary embolism;
    * myocardial infarction;
    * severe or unstable arrhythmia or angina;
    * percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting;
    * Cerebrovascular accident, transient ischemic attack, and cerebral embolism.
* Have received a stem cell transplant or an organ transplant.
* Patients who need to use during the study or have used or the following drugs within 14 days prior to the first dose: CYP3A4 strong inhibitor or strong inducer; warfarin or any other coumarin derivative anticoagulant.
* The investigator judges other severe, acute or chronic medical illness or laboratory abnormalities that may increase the risk associated with the study or may interfere with the interpretation of the findings.
* The investigator judged that the patient's compliance was poor or that there were other conditions that were not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate according to RECIST 1.1 | 12 months
  The proportion of patients with complete remission (CR) and partial remission (PR) in all patients.Disease progression will be evaluated according to RECIST 1.1.

SECONDARY OUTCOMES:
Disease Control Rate according to RECIST 1.1 and iRECIST | 12 months
  The proportion of patients with complete remission (CR),partial remission (PR) and stable disease(SD) in all patients.Disease progression will be evaluated according to RECIST 1.1 and iRECIST.
Duration of Response according to RECIST 1.1 and iRECIST | 12 months
  The time interval between the first time of being evaluated as complete response (CR) or partial response (PR) and the first time of being evaluated as progressed disease(PD). Disease progression will be evaluated according to RECIST 1.1 and iRECIST.
Time to Response to RECIST 1.1 and iRECIST | 12 months
  Time from randomization to complete response (CR) or partial response (PR). Disease progression will be evaluated according to RECIST 1.1 and iRECIST
Progression-free survival | 12 months
  The internal between the date of randomization and the date of disease progression, unaccepted toxicity, or death.
Overall survival | 36 months
  The internal between the date of randomization and the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Jun, M.D, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China